CLINICAL TRIAL: NCT03608930
Title: Comparison of Hot Snare Polypectomy Using Regular or Rotary Polypectomy Snare for the Resection of Colorectal Polyps: a Prospective Randomized Controlled Trial
Brief Title: Comparison of Using Regular or Rotary Polypectomy Snare for the Resection of Colorectal Polyps
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ningbo No. 1 Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RSCP2018-V1.0
Record Dates: First submitted 2018-07-12; First posted 2018-08-01 (Actual); Last update posted 2019-07-02 (Actual); Status verified 2018-07

CONDITIONS: Polypectomy Snare

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- rotary polypectomy snare (Experimental): All colorectal polyps found are removed using a rotary polypectomy snare (Disposable Polypectomy Snare). The technique is hot snare resection of the polyp with electrocautery. Details are as follows: (1) insert the snare into the colonoscopy; (2) connect the snare with the high-frequency device;(3) advance sliding handle to open the loop; (4) adjust the direction of the snare by rotating the handle as required, rotate the loop until the loop reaches target polyp; (6) encircle the target polyp with loop; (7) pull the sliding handle, lasso the target polyp;(8) resect the polyp with electrocautery, then inhaling the transected polyp into a trap followed by submission to the histological evaluation. The hemostatic clipping is used after hot snare polypectomy if removing a flat polyp or bleeding on the wound after treatment.
  Interventions: Device: Disposable Polypectomy Snare,JHY-SD-23-230-30-A1
- regular polypectomy snare (No Intervention): All colorectal polyps found are removed using a regular polypectomy snare (polypectomy snare, symmetrical). The technique is hot snare resection of the polyp with electrocautery. Details are as follows: (1) insert the snare into the colonoscopy; (2) connect the snare with the high-frequency device;(3) advance sliding handle to open the loop; (4) adjust the bending section angulation of the colonoscopy as required, advance the snare until the loop reaches target polyp; (6) encircle the target polyp with loop; (7) pull the sliding handle, lasso the target polyp;(8) resect the polyp with electrocautery, then suction of the transected polyp into a trap followed by submission to the histological evaluation. The hemostatic clipping is performed after hot snare polypectomy if a flat polyp or bleeding on the wound after treatment.

INTERVENTIONS:
Device: Disposable Polypectomy Snare,JHY-SD-23-230-30-A1 — The technique is hot snare resection of the polyp with electrocautery. Details are as follows: (1) insert the snare into the colonoscopy; (2) connect the snare with the high-frequency device;(3) advance sliding handle to open the loop; (4) adjust the direction of the snare by rotating the handle as required, rotate the loop until the loop reaches target polyp; (6) encircle the target polyp with loop; (7) pull the sliding handle, lasso the target polyp;(8) resect the polyp with electrocautery, then inhaling the transected polyp into a trap followed by submission to the histological evaluation.
  Arms: rotary polypectomy snare

SUMMARY:
This clinical trial is being conducted to assess whether the rotary polypectomy snare could decrease the time to removal of colorectal polyps

ELIGIBILITY:
Inclusion Criteria:

18-85 year;

Patients with colorectal polyps ;

informed consent;

Exclusion Criteria:

patients taking antiplatelet or anticoagulant therapy during the past 1 week of the procedure;

known coagulopathy;

history of inﬂammatory bowel diseases;

Hemodynamically unstable;

pregnancy

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2018-08-01 (Actual); Primary Completion 2018-08-02 (Actual); Study Completion 2018-09-30 (Actual)

PRIMARY OUTCOMES:
the average time of each polyp removing | 1day
  Using a stopwatch to record the removing time of each polyp (starting the stopwatch when the snare stretched out of the pipe and ending with the polyp being completely removed); Furthermore, we excluded the time of submucosal injection, electrocoagulation, and the use of preventive titanium clips

SECONDARY OUTCOMES:
Postpolypectomy bleeding | 2 weeks
  Postpolypectomy bleeding within two weeks after polypectomy

OTHER OUTCOMES:
The procedure time | 1day
  The procedure time spent for polypectomy

CONTACTS AND LOCATIONS:
Overall Officials: Lei XU, PHD, Principal Investigator — Department of Gastroenterology, Ningbo No. 1 Hospital, Ningbo, China
Locations (1):
- Ningbo NO.1 hospital, Ningbo, Zhejiang, China

IPD SHARING:
Plan to Share IPD: Undecided